CLINICAL TRIAL: NCT06612073
Title: Evaluation Of The Degree Of Kidney Injury in Children With Hypovolemic Shock
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Tarek Mohamed Mahmoud, Doctor, Assiut University
Other Study IDs: AKI with hypovolemic shock
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Evaluation of Acuty Kidney Injury in Children With Hypovolemic Shock
Keywords: AKI in hypovolemic shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children who have kidney affection after hypovolemic shock: No intervtional drugs or devices at all.

SUMMARY:
To evaluate renal affection and its degree in hypovolemic shocked

children

DETAILED DESCRIPTION:
Acute kidney injury is a syndrome characterised by the rapid loss of the kidney's excretory function and is typically diagnosed by the accumulation of end products of nitrogen metabolism (urea and creatinine) or decreased urine output, or both. It is the clinical manifestation of several disorders that affect the kidney acutely. Acute kidney injury is common in hospital patients and very common in critically ill patients. In these patients, it is most often secondary to extrarenal events.. In low-income and middle-income countries, infections and hypovolaemic shock are the predominant causes of AKI. In high-income countries, AKI mostly occurs in elderly patients who are in hospital, and is related to sepsis, drugs or invasive procedures. Infection and trauma-related AKI and AKD are frequent in all regions.

There are numerous potential causes of AKI, mainly related to a focal mismatch between oxygen and nutrient delivery (because of impaired microcirculation) to the nephrons and increased energy demands (due to cellular stress).

The prerenal form of AKI is due to any cause of reduced blood flow to the kidney. This may be part of systemic hypoperfusion resulting from hypovolemia or due to selective hypoperfusion of the kidneys, such as

* Hypovolemia: hemorrhage, severe burns, and gastrointestinal fluid losses such as diarrhea, vomiting, and high ostomy output.
* Hypotension from systemic vasodilation: septic shock, anaphylaxis, anesthesia administration.
* Glomerular efferent arteriolar vasodilation (causing intraglomerular hypotension): ACE inhibitors, angiotensin receptor blockers.

Diagnosis

• Increase in serum creatinine by 0.3 mg/dL or more (26.5 μmol/L or more) within 48 hours And other diagnostic criteria according to the stage Shock is the state of insufficient blood flow to the tissues of the body as a result of problems with the circulatory system.[5][6]Initial symptoms of shock may include weakness, fast heart rate, fast breathing, sweating, anxiety, and increased thirst Shock is divided into four main types based on the underlying cause: hypovolemic, cardiogenic, obstructive, and distributive shock.Hypovolemic shock, also known as low volume shock, may be from bleeding, diarrhea, or vomiting.

One of most common complication of shock is acute kidney injury due to decrease perfusion to kidney which can improved once shock improved

Management :

Aggressive intravenous fluids are recommended in most types of shock (e.g. 1-2 liter normal saline bolus over 10 minutes or 20 mL/kg in a child) which is usually instituted as the person is being further evaluated.[7] Colloids and crystalloids appear to be equally effective with respect to outcomes.,[8] Balanced crystalloids and normal saline also appear to be equally effective in critically ill patients.[9] If the person remains in shock after initial resuscitation, packed red blood cells should be administered to keep the hemoglobin greater than 100 g/L.

Some AKI patients tend to develop volume overload, which should be corrected as early as possible to avoid pulmonary and cardiac complications. Euvolemic state can be achieved with the help of diuretics, which is a cornerstone in managing such patients. Usually, high doses of IV furosemide are needed to correct volume overload in AKI patients; however, it plays no role in converting oliguric AKI to non-oliguric AKI.

In some cases, short-term renal replacement therapy is needed for AKI until the kidney function recovers. Some indications for RRT are severe and non-responsive hyperkalaemia, uremic pericarditis, and pulmonary oedema where the patient is prone to develop multiple electrolyte and acid-base abnormalities as well as fluid overload.

Dialysis in this setting is usually performed through a temporary venous catheter when required. Continuous renal replacement therapy can also be utilized in patients who cannot tolerate haemodialysis due to hypotension. It is a much slower, continuous type of dialysis. . Metabolic acidosis is one such instance where systemic administration of citrate or bicarbonate is often required to maintain a suitable blood pH. The requirement for renal replacement therapy should be re-evaluated daily. Renal replacement therapy is usually required for short periods, ranging from a few days to a few weeks; however, some cases can take months to recover and may require intermittent RRT support.

ELIGIBILITY:
Inclusion Criteria:

Patient with hypovolemic shock affecting kidney function below 18 Years' old.

Exclusion Criteria:

* Patients with kidney function affection due to any type of shock other

Than hypovolemic shock .

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: It is aprospective cohort study to detect acute kidney injury after hypovolemic shock in children from age 1 day till 18 years to help in minimize risk factor .
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of renal affection and its degree in patient with hypovolemic shock | Baseline
  Detect patient with kidney affection (raised urea ,creatinine and electrolyte)

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uchino S, Bellomo R, Goldsmith D, Bates S, Ronco C. An assessment of the RIFLE criteria for acute renal failure in hospitalized patients. Crit Care Med. 2006 Jul;34(7):1913-7. doi: 10.1097/01.CCM.0000224227.70642.4F. PMID 16715038
- [Result] Hegarty NJ, Young LS, Kirwan CN, O'Neill AJ, Bouchier-Hayes DM, Sweeney P, Watson RW, Fitzpatrick JM. Nitric oxide in unilateral ureteral obstruction: effect on regional renal blood flow. Kidney Int. 2001 Mar;59(3):1059-65. doi: 10.1046/j.1523-1755.2001.0590031059.x. PMID 11231361
- [Result] Kellum JA, Romagnani P, Ashuntantang G, Ronco C, Zarbock A, Anders HJ. Acute kidney injury. Nat Rev Dis Primers. 2021 Jul 15;7(1):52. doi: 10.1038/s41572-021-00284-z. PMID 34267223
- See also: Related Info — https://nephrologypc.com/